CLINICAL TRIAL: NCT06017167
Title: Dexmedetomidine Versus Dexamethasone Adding to Ondansetron for Prophylaxis Against Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy
Brief Title: Prophylaxis Against Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, yasmine mohammed mahmoud mustafa eldeba, Resident doctor of Anaesthesia and ICU Department, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PONV after lap cholecystectomy
Record Dates: First submitted 2023-08-14; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Nausea and Vomiting; Laparoscopic Cholecystectomy
Keywords: dexamethasone; dexmedetomidine; ondansetron
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron; Dexmedetomidine; Saline Solution; halofantrine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients will be randomly classified with computer generated random numbers into two equal groups (each group 35 patients) Group I: will receive Ondansetron 4mg + dexmedetomidine 0.5 ug/kg + normal saline to complete 10 ml. volume IV infusion over 10 minutes.
  Group II: will receive Ondansetron 4mg + dexamethasone 8mg + normal saline to complete 10 ml volume IV ifusion over 10 minutes.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
  * The participants will be kept blind in both groups.
  * Outcome assessors will be blinded as they will be anesthesia resident and nurse not participating in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Active Comparator): will receive ondansetron 4mg + dexmedetomidine 0.5 ug/kg + normal saline to complete 10 ml. volume IV infusion over 10 minutes.
  Interventions: Drug: Ondansetron 4mg + dexmedetomidine 0.5 ug/kg + normal saline .
- Dexamethasone Group (Active Comparator): will receive Ondansetron 4mg + dexamethasone 8mg + normal saline to complete 10 ml. volume IV infusion over 10 minutes.
  Interventions: Drug: Ondansetron 4mg + dexamethasone 8mg + normal saline.

INTERVENTIONS:
Drug: Ondansetron 4mg + dexmedetomidine 0.5 ug/kg + normal saline . — compare antiemetic effects between dexmedetomidine and ondansetron in the first group versus dexamethasone and ondansetron in the second group
  Other Names: ondansetron 4mg (Zofran; GlaxoSmithKline, Alexandria, USA; dexmedetomidine (Precedex; Ho-Spira Inc., Lake Forest, Illinois, USA
  Arms: Dexmedetomidine Group
Drug: Ondansetron 4mg + dexamethasone 8mg + normal saline. — Group II: Ondansetron 4mg + dexamethasone 8mg + normal saline.
  Other Names: ondansetron 4mg (Zofran; GlaxoSmithKline, Alexandria, USA; dexamethasone; Amriya Pharmaceutical Industries, Egypt
  Arms: Dexamethasone Group

SUMMARY:
The aim of the study is to compare antiemetic effects between dexmedetomidine and ondansteron in the first group versus dexamethasone and ondansteron in the second group.

The primary outcome in this study is incidence of postoperative nausea and vomiting after laparoscopic cholecystectomy.

The secondary outcomes are:

* The severity of post operative nausea and vomiting.
* Use of rescue antiemetic drugs.
* Postoperative pain and sedation.

DETAILED DESCRIPTION:
General anesthesia is widely used in several surgeries. It can cause some complications such as postoperative nausea and vomiting (PONV). PONV is more common in general anesthesia than spinal anesthesia. PONV remains an extremely significant challenge due to its complex mechanism, resulting in serious consequences. Therefore an effective way to prevent or arrest PONV is urgently needed as Also, it can cause electrolyte imbalance and aggravate bleeding that delay hospital discharge.

The causes of PONV are multifactorial and can largely be categorized as patient risk factors, anaesthetic technique, and surgical procedure. Antiemetics work on several different receptor sites to prevent or treat PONV.

No single antiemetic pharmaceutical has been provided to be a universal solution to PONV. In general, multimodal combination treatment has superior viability for PONV prophylaxis compared with monotherapy .

Because nausea and vomiting were defined as two separate phe-nomena, studies should report and evaluate the variables distinctly . While since few patients experience vomiting without nausea, the incidence of PONV and postoperative nau¬sea (PON) is fairly similar, thus original papers often do not try to distinguish these variables . So, if PONV but not PON was reported in trails, we considered the PONV variables as a very close substitute for PON; when both PONV and PON were reported simultaneously, we assessed the nausea values. The most com¬monly used time interval to measure the role of antiemetic is 24 hours 6.

Ondansetron is a serotonin receptor antagonist, which is very important in preventing nausea and vomiting due to surgery and chemotherapy; it exhibited an anti-vomiting effect by inhibiting 5-Hydroxytryptamine type 3 (5-HT3) receptors in the vomiting centre .

Dexmedetomidine is a potent and highly selective a2-adrenoceptor agonist, which binds to transmembrane G protein-binding receptor located in the brain and spinal cord. Since nausea and vomit¬ing may be induced by high catecholamine con¬centrations, a decrease of sympathetic tone could explain the antiemetic effect of dexme¬detomidine. Finally, consumption of intraopera¬tive opioids, which increases the risk of PONV , may be reduced through the use of dexmedetomidine It affects the functions of central nervous, circulatory systems and exhibits sedative, analgesic, sympatholytic properties. Recently, the effect of dexmedetomidine on PONV has been the focus of clinical researchers. Nevertheless, controversy about the effectiveness of dexmedetomidine for PONV is still ongoing, for different results reported in associated literature.

Glucocorticoids may exert an antiemetic effect by inhibiting inflammatory mediators and by interacting with serotonin, neurokinin, a-adrenergic receptors, and other receptors. Furthermore, several studies have shown that dexamethasone enhances the antiemetic efficacies of 5-hydroxytryptamine type 3 (5-HT3) receptor antagonists.

ELIGIBILITY:
Inclusion Criteria:

* 70 Female patients aged between 18 and 65 years
* ASA I or II
* patients scheduled for elective laparoscopic cholecystectomy surgery will be included in this study.

Exclusion Criteria:

* Females above 65 years old.
* patients under 18 years old.
* ASA > II.
* Obesity (BMI>40 kgm2).
* Known hypersensitivity to drugs used in the study protocol.
* Comorbidities that were known to increase the risk of PONV (e.g. vestibular disease).
* Liver or renal dysfunction (liver enzyme or creatinine 1.5 times higher than normal).
* Alcoholism or drug abuse.
* Use of antiemetics and psychotropic drugs or glucocorticoids within 24 h before surgery.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — According to APFEL score female is a risk factor for PONV.
Enrollment: 70 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative nausea and vomiting after laparoscopic cholecystectomy. | through out 24 hours after surgery.
  The incidence of vomiting, use of rescue antiemetics, and analgesic requirements were recorded at 0 to 1 hours after surgery in the postanesthetic care unit (PACU)At 6 and 24 hours after surgery, the incidence and severity of PONV were assessed using the Rhodes Index of nausea, vomiting, and retching.

SECONDARY OUTCOMES:
The severity of post operative nausea and vomiting. | During 24 hours after surgery.
  The severity of nausea was evaluated using a 10-point numerical rating scale (NRS) At 6 and 24 hours after surgery, the incidence and severity of PONV were assessed using the Rhodes Index of nausea, vomiting, and reteching.At 6 and 24 hours after surgery.
  The Rhodes Index is a reliable and valid patient self-reporting tool to assess nausea, vomiting, and retching and consists of eight items with 5 scales (0-4). This index has been shown to be a highly reliable method for evaluating gastrointestinal distress after ambulatory surgery.
- Postoperative pain | During 24 hours after surgery.
  Pain score was also assessed using a 10-point NRS.
- Postoperative sedation | During 24 hours after surgery.
  Ramsay sedation score (1=agitated, anxious, or restless; 2=oriented, cooperated, and tranquil; 3=responsive to verbal commands only; 4=asleep, brisk response to a loud auditory stimulus or a light glabella tap; 5=sluggish response to a glabella tap or loud auditory stimulus; 6=no response to a loud auditory stimulus or a light glabella tap) were recorded. Over-sedation was defined as a Ramsay sedation score>4.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Lotfy, PHD, Principal Investigator — Assistant Professor of Anesthesia and Intensive Care, Tanta Univ
Locations (1):
- Tanta University hospitals, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available with the principle investigator within 6 months after publishing the study
Supporting Information: Study Protocol, SAP
Time Frame: within 6 months after publishing the study
Access Criteria: yasmine162078_pg@med.tanta.edu.eg

REFERENCES:
- [Background] Rhodes VA, McDaniel RW. The Index of Nausea, Vomiting, and Retching: a new format of the lndex of Nausea and Vomiting. Oncol Nurs Forum. 1999 Jun;26(5):889-94. PMID 10382187